CLINICAL TRIAL: NCT04451746
Title: The Influence of Combined Oral Contraception on the DEvelopment and progRession of Chronic venoUs diSeases
Acronym: ICODERUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinic of Phlebology and Laser Surgery, Chelyabinsk, Russia (Other)
Responsible Party: Principal Investigator, Denis Borsuk, Clinic of Phlebology and Laser Surgery, Clinic of Phlebology and Laser Surgery, Chelyabinsk, Russia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 000000114
Record Dates: First submitted 2020-06-24; First posted 2020-06-30 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Chronic Venous Diseases
MeSH Terms: interventions — Contraceptives, Oral, Combined

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tableted hormonal drugs for contraception (Other): Tableted hormonal drugs for contraception, 1) COCs with bioidentical estrogen; 2) COCs with ethinyl estradiol 30mkg according to the scheme 21 + 7; 3) COCs with ethinyl estradiol 20mkg according to the scheme 21 + 7.
  Interventions: Drug: Combined Oral Contraceptive

INTERVENTIONS:
Drug: Combined Oral Contraceptive — The investigators consistently include patients who have been prescribed hormonal tablets for contraception, namely 1) COCs with bioidentical estrogen; 2) COCs with ethinyl estradiol 30mkg according to the scheme 21 + 7; 3) COCs with ethinyl estradiol 20mkg according to the scheme 21 + 7.

SUMMARY:
Investigation of the influence of combined oral contraception on the development and progression of chronic venous diseases

ELIGIBILITY:
Inclusion Criteria:

1. The investigators consistently include patients who have been prescribed hormonal tablets for contraception, namely 1) COCs with bioidentical estrogen; 2) COCs with ethinyl estradiol 30mkg according to the scheme 21 + 7; 3) COCs with ethinyl estradiol 20mkg according to the scheme 21 + 7.
2. Clinical class C0-1 according to CEAP;

2) Able to come for checkups every 3 months; 3) The presence of informed consent.

Exclusion Criteria:

1. Age up to 45 years;
2. A history of surgical treatment of veins of the lower extremities;
3. Clinical class C2 and higher according to CEAP;
4. History of DVT or PE;
5. Aplasia or angio-dysplasia of deep veins;
6. Restriction of mobility;
7. Arterial insufficiency;
8. Oncological diseases.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-24 (Actual); Primary Completion 2025-07-24 (Estimated); Study Completion 2025-08-24 (Estimated)

PRIMARY OUTCOMES:
Development and progression of chronic venous diseases | 1 year

SECONDARY OUTCOMES:
Deep venous thrombosis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Fokin, Study Chair — South Ural State Medical University
Locations (1):
- Clinic of phlebology and laser surgery, Chelyabinsk, Russia

IPD SHARING:
Plan to Share IPD: Undecided